CLINICAL TRIAL: NCT03223636
Title: Measuring the Latency Connectome in the Central Nervous System Using Neuroimaging and Neurophysiological Techniques
Brief Title: Measuring the Latency Connectome in the Central Nervous Systems Using Neuroimaging and Neurophysiological Techniques
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170128; 17-N-0128
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
Keywords: Transcranial Magnetic Stimulation (TMS); Magnetic Resonance Imaging (MRI); Electroencephalogram (EEG); Magnetoencephalogram; Transcranial Electrical Stimulation (TES)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers
  Interventions: Device: TMS; Device: MRI

INTERVENTIONS:
Device: TMS — We will use TMS with paired-pulse technique to activate corticospinal neurons in the primary motor cortex and motorneurons in the brainstem, respectively (Hallett 2007; Ugawa et al. 1991; Ugawa et al.1994). Two stimulations will be separated with various interstimulus intervals to produce collision on nerve fibers with different conduction velocity in the corticospinal tract. The conduction time on nerve fibers in the corticospinal tract with different conduction velocity will be identified and the distribution of these fibers will be calculated.
Device: MRI — MRI exams will consist of several sessions including calibration, anatomic, and diffusion MRI scanning (Avram et al. 2013; Avram et al. 2016; Pierpaoli et al. 1996). Data in each exam will be acquired in the left or right forearm (PNS).

SUMMARY:
Background:

Little is known about the time it takes for nerve signals to go from one area of the brain to another. Using advanced methods for brain research, researchers want to look at the time it takes to send messages between different brain areas. They also want to develop new tests.

Objectives:

To develop tests to measure the sizes of nerve fibers in the peripheral nerve system and in the brain. Also to find out the different speeds that information travels in nerve fibers.

Eligibility:

Healthy, right-handed people ages 18-70

Design:

Participants will be screened with medical history and a physical exam.

Participants will have up to 7 visits depending on the tests they choose. Visits last about 2-4 hours and may involve the following tests:

* Physical exam
* Urine tests
* Magnetic resonance imaging (MRI). Participants lie on a table that slides into a scanner. They will be in the scanner for up to 1 hour. For some scans, sensors are placed on the skin. They will get earplugs for loud noises.
* Small, sticky pads on the skin will electrically stimulate nerves in the forearm.
* Transcranial magnetic stimulation (TMS). A wire coil will be held to the scalp. A brief electrical current passes through the coil to affect brain activity.
* Electroencephalography. TMS will be given to the brain. Small electrodes on the scalp measure brain activity. Participants may do small tasks.
* Electrodes on the scalp will send an electrical current to the brain.
* A cone with magnetic detectors will be lowered onto the head to record brain activity. Participants will perform various tasks.

DETAILED DESCRIPTION:
Objectives:

We are proposing the development and assessment of an MRI and neurophysiology-based experimental and theoretical framework to measure peripheral and intercortical latencies and latency distributions in the living human. This entails combining and integrating neurophysiological and neuroimaging so that we can eventually generate latency and latency distribution matrices for central nervous systems (CNS) using neuroimaging techniques. Neuroimaging and neurophysiological studies in the peripheral nerve system (PNS) will provide essential data for proof-of-concept and for validating this approach.

Study Population:

We intend to study up to 40 healthy volunteers. Each subject will complete 1 to 8 visits involving various measurements with different neuroimaging and neurophysiological techniques.

Design:

This is an exploratory study that consists of different measurements using multimodal neurophysiological and neuroimaging techniques. Diffusion magnetic resonance imaging (MRI), mean apparent propagator (MAP)-MRI, AxCaliber MRI, multiple pulsed field gradient MRI, and resting-state functional MRI will be performed in 1 to 2 visits. In another 1 to 5 visits, we will use neurophysiological techniques including peripheral electrical stimulation, transcranial magnetic stimulation (TMS), electroencephalography (EEG) and magnetoencephalography (MEG) with various experimental paradigms to correlate with the latency and latency distribution matrices generated by neuroimaging techniques. All these techniques are exploratory and success or failure of one of them does not have immediate implications for the others.

Outcome Measures:

We will measure average axon diameter (AAD) and axon diameter distributions (ADD), as well as compute white matter pathway trajectories using diffusion MRI and MAP-MRI data, and use resting-state functional MRI to measure blood oxygenation level-dependent signal to identify salient cortical regions in which many of these tracts terminate. For proof-of-concept measurements in the PNS, compound muscle action potential or surface compound nerve action potential on the skin will be measured following peripheral nerve stimulation. For TMS , we will measure motor evoked potential (MEP) amplitude. Cortical evoked potential in different cortical areas induced by TMS will be measured in EEG recordings. We will study millisecond coupling delays between different cortical areas with MEG. We will measure time and phase delays as computed from whole-head signals in the subject. Coherence analysis for cortical activity with EEG and MEG recordings between different cortical areas will be performed. We will attempt to correlate MRI measurements with the individual physiological measurements.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ages between 18-70 years.
* Right-handed (tested by the Edinburg handedness inventory).
* Able to give informed consent and able to comply with all study procedures.

EXCLUSION CRITERIA:

* Self-reported consumption of >14 alcoholic drinks/week for a man and >7 alcoholic drinks/week for a woman.
* Abnormal findings on neurological examination.
* History of brain tumor, stroke, head trauma with loss of consciousness, epilepsy or seizures.
* Current episode of any major psychiatric illness.
* Use of medications that act directly on the CNS.
* Hearing loss reported in the history or detected in the routine physical examination
* Having permanent tattooed makeup (eyeliner, lip, etc.) or general tattoos. Subjects with tattoos will be excluded if those are in a dangerous location in the body or made with colors (e.g. dark blue and dark green) whose content in iron cannot be definitely ruled out by the investigators.
* Having non-organic implant or any other device such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch, any metallic implants or objects, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunt.
* Having cerebral or other aneurysm clips.
* Having shrapnel or other metal imbedded in the body (such as from war wounds or accidents).
* Had severe accidents in the past that may possibly have left metal in the body.
* Previously worked in metal fields or with machines that may have left any metallic fragments in or near eyes.
* Having any psychological contraindications for MRI (e.g., suffer from claustrophobia, unable to lie comfortably on your back for 2 hours).
* Discomfort being in a small space for the expected length of the experiment, up to 2 hours.
* Pregnancy.
* NIH staff from HMCS in NINDS, Section on Quantitative Imaging and Tissue Sciences in NICHD or MEG Core facility in NIMH involved in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
measure motor evoked potential (MEP) amplitude | throughout
  For TMS, we will measure motor evoked potential (MEP) amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Ni Z, Leodori G, Vial F, Zhang Y, Avram AV, Pajevic S, Basser PJ, Hallett M. Measuring latency distribution of transcallosal fibers using transcranial magnetic stimulation. Brain Stimul. 2020 Sep-Oct;13(5):1453-1460. doi: 10.1016/j.brs.2020.08.004. Epub 2020 Aug 11. PMID 32791313
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-N-0128.html